CLINICAL TRIAL: NCT07168512
Title: "Myofascial Release With or Without Exercise for Cervicogenic Headache"
Brief Title: Effect of Myofascial Release Technique Alone or Combined With Exercises on Cervical Cobb Angle, Sleep Quality, and Psychological Factors in Patients With Cervicogenic Headache
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mosab ALdabbas, mosab aldabbas, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Al Azhar university, Palestine
Record Dates: First submitted 2025-08-27; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Effect of Physiotherapy on Cobb Angle in Patients With Cervicogenic Headache
Keywords: cobb angle; sleep; cervicogenic headache; exercise; myofascial release
MeSH Terms: conditions — Post-Traumatic Headache; Motor Activity | interventions — Exercise; Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- One group will receive exercises (Experimental): The intervention will include targeted neck strengthening and endurance exercises combined with the application of hot packs
  Interventions: Other: Exercises (Endurance and strengthening)
- Exercises and Myofascial release technique (Experimental): The intervention will include targeted neck strengthening and endurance exercises combined with the application of hot packs in addition to myofasical release technique
  Interventions: Other: Exercises (Endurance and strengthening); Other: Myofascial release technique
- Control (No Intervention): control ; only advices

INTERVENTIONS:
Other: Exercises (Endurance and strengthening) — Neck Strengthening and Endurance Exercises with Hot Packs
  Preparation: A moist hot pack will be applied for 10-15 minutes to the cervical region before exercise to reduce stiffness and enhance tissue extensibility.
  Exercise program:
  Deep cervical flexor training: Chin tucks in supine and sitting, progressing to sustained isometric holds.
  Extensor and scapular stabilizer training: Prone head lifts and shoulder retraction exercises with light resistance.
  Endurance training: Low-load, high-repetition exercises focusing on maintaining cervical posture against gravity.
  Progression: Intensity and duration will gradually increase, emphasizing endurance over maximal strength to correct postural deficits.
  Frequency: 40 minutes per session, 3 times per week for 6 weeks
  Rationale: The combined use of heat and targeted exercises improves neuromuscular control, enhances cervical stability, and supports better cervical curvature correction. Myofascial Release Technique
  Arms: Exercises and Myofascial release technique; One group will receive exercises
Other: Myofascial release technique — Myofascial Release Technique
  Target areas: Suboccipital muscles, upper trapezius, levator scapulae, and deep cervical fascia.
  Method: A physiotherapist will perform gentle, sustained manual pressure and low-load, long-duration stretching on restricted cervical and upper thoracic fascia to reduce tension and improve soft tissue mobility.
  Duration and frequency: Each session will include 30'to 50 minutes of myofascial release, delivered 3 times per week for the study period for 6 weeks.
  Rationale: This technique aims to decrease myofascial restrictions contributing to abnormal cervical alignment and pain, thereby facilitating improved posture and muscle activation.
  Arms: Exercises and Myofascial release technique

SUMMARY:
This study will investigate whether myofascial release therapy alone or in combination with therapeutic exercises can improve cervical spine alignment, measured by cervical Cobb angle on X-ray, in patients with cervicogenic headache. The research will also examine potential effects on sleep quality and psychological factors."

ELIGIBILITY:
Inclusion Criteria:

* Age 20-55 years.
* Clinical diagnosis of cervicogenic headache according to International Classification of Headache Disorders (ICHD-3) criteria (headache attributed to cervical disorder).

Exclusion Criteria:

* History of major cervical spine pathology such as fracture, dislocation, congenital malformation, tumor, infection, or inflammatory arthritis (e.g., rheumatoid arthritis, ankylosing spondylitis).
* Previous cervical spine surgery or fusion at any level.
* Red flag symptoms indicating serious pathology (e.g., progressive neurological deficit, unexplained weight loss, fever, history of cancer).
* Systemic or neurological disorders that may affect neck function or headache (e.g., multiple sclerosis, Parkinson's disease).
* Severe osteoporosis or metabolic bone disease that contraindicates cervical X-ray imaging.
* Vascular disorders such as vertebrobasilar insufficiency or carotid artery disease.
* Pregnancy or breastfeeding (due to radiation exposure during cervical radiography).
* Unstable psychiatric conditions (e.g., severe depression, psychosis) that may interfere with participation or adherence.
* Recent physiotherapy or manual therapy targeting the cervical region within the past 6 weeks, or planned during the study outside the protocol.
* Use of botulinum toxin or steroid injections to the neck or head region in the past 6 months.
* Contraindications to manual therapy or exercise (e.g., acute cervical disc herniation, severe myelopathy, unstable cardiovascular disease).
* Inability to understand study procedures, comply with treatment sessions, or provide informed consent.
* Symptoms of migraine, tension-type headache (TTH), or any other headache apart from cervicogenic headache.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-04 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-03 (Estimated)

PRIMARY OUTCOMES:
Cervical cobb angle | pre and post (6 weeks)
Cobb angle of cervical spine assessed by X Ray (Lateral) | pre , and 8 weeks post physiotherapy intervention
  Landmarks & angle construction (C2-C7 Cobb)
  Draw a line along the inferior endplate of C2.
  Draw a line along the inferior endplate of C7.
  Erect perpendiculars to each line and measure the angle at their intersection (alternatively, measure the acute angle between the two endplate lines and subtract from 180°).
  Record the angle in degrees of lordosis (greater positive values = greater lordosis). Note the sign convention in your CRF and keep it consistent pre/post.
  Normal value is between 20_40
Hospital Anxiety and depression scale | pre and 8 weeks post physiotherapy interventions
  The Hospital Anxiety and Depression Scale (HADS) is a validated self-report screening tool developed to assess levels of anxiety and depression in patients, particularly in non-psychiatric hospital settings. It contains 14 items divided into two subscales: seven items for anxiety (HADS-A) and seven for depression (HADS-D). Each item is scored on a 4-point Likert scale ranging from 0 to 3, giving a maximum score of 21 for each subscale. Higher scores indicate greater symptom severity. Scores of 0-7 are generally considered normal, 8-10 suggest borderline (possible) anxiety or depression, and 11-21 indicate clinically significant levels. The HADS is widely used in clinical and research contexts due to its brevity, ease of administration, and ability to distinguish between anxiety and depression symptoms without being confounded by physical illness.

SECONDARY OUTCOMES:
sleep quality | pre, and 8 weeks post physiotherapy
  The Pittsburgh Sleep Quality Index (PSQI) is a widely used self-report questionnaire designed to assess sleep quality and disturbances over a one-month period. It consists of 19 items grouped into seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Each component is scored from 0 (no difficulty) to 3 (severe difficulty), and the component scores are summed to yield a global score ranging from 0 to 21. A higher score indicates poorer sleep quality, with a global score greater than 5 commonly used to differentiate between good and poor sleepers. The PSQI is valued for its reliability, validity, and practicality in both clinical and research settings for evaluating sleep problems across diverse populations.
neck disability | pre and 8 weeks post physiotherapy interventions
  The Neck Disability Index (NDI) is a self-administered questionnaire designed to measure a patient's level of neck pain-related disability. It consists of 10 items covering domains such as pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreation. Each item is scored on a 6-point scale ranging from 0 (no disability) to 5 (complete disability), resulting in a total possible score of 50. The raw score is often expressed as a percentage by multiplying by two. Higher scores indicate greater disability, with common interpretation ranges being: 0-4 (no disability), 5-14 (mild), 15-24 (moderate), 25-34 (severe), and ≥35 (complete disability). The NDI is one of the most widely used tools for assessing functional status in patients with neck pain, demonstrating strong reliability, validity, and responsiveness to clinical change.

CONTACTS AND LOCATIONS:
Locations (2):
- Palestinian Territories (2):
  - Naser Medical Complex, Gaza, Gaza Strip
  - Ministry of Health, Gaza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cervical Cobb angle, sleep quality and psychological factors in patients with chronic neck pain with and without cervicogenic headache
- See also: Related Info — https://sheets.new